CLINICAL TRIAL: NCT00347308
Title: Photographic Assessment of Eyebrow Position and Range of Motion
Status: Completed | Type: Observational
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Anthony P. Sclafani, Director of Facial Plastic Surgery, The New York Eye & Ear Infirmary
Other Study IDs: 001
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-04

CONDITIONS: Brow Ptosis
Keywords: brow ptosis, facial aesthetics, browlift, facelift

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Eyebrow Position — Photography of brow positions

SUMMARY:
Forehead and eyebrow surgery is a frequently performed cosmetic surgical procedure in which the eyebrows are raised to a more aesthetically pleasing position. Typically, this position is judged by the surgeon pre-operatively based on traditional aesthetic concepts, some of which date to the Classical era. This study is designed to assess the variance of the eyebrow from the desired aesthetic position (as determined by the subject), as wel as to assess the distance of normal excursion of the brow from maximum voluntary depression to maximum voluntary elevation.

DETAILED DESCRIPTION:
A set of 5 digital photographs will be taken of 100 (30 male, 70 female) adult study participants. Prior to photography, water soluble ink will be used to mark the inferior aspect of the superior orbital rim above the medial and lateral canthi and in the mid pupillary line. Photographs taken will image patients from crown to chin and will be taken with eyes open and closed, brows raised, maximally contracted and at rest. A final photograph will be taken with the subject manually holding both brows in the position he/she finds most aesthetically pleasing as seen in a mirror. During all photography, a ruler will be held against the face for later calibration, all photographs will be taken with a camera mounted flash and with the patient in a Frankfort horizontal plane. All photographs will be analyzed with proprietary computer software.

ELIGIBILITY:
Inclusion Criteria:

* adults,
* aged 18-85 years

Exclusion Criteria:

* prior forehead, eyebrow or eyelid surgery,
* neurotoxin treatment to the forehead or eyes within the past 6 months,
* injectable soft tissue filler used within the last 12 months,
* photosensitivity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, between the ages of 18- 85
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sclafani, MD, Principal Investigator — The New York Eye & Ear Infirmary
Locations (1):
- Center for Facial Plastic Surgery, Chappaqua, New York, United States

REFERENCES:
- [Derived] Sclafani AP, Jung M. Desired position, shape, and dynamic range of the normal adult eyebrow. Arch Facial Plast Surg. 2010 Mar-Apr;12(2):123-7. doi: 10.1001/archfacial.2010.17. PMID 20231595

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: All patients entered into the study
Period: Overall Study
Arm/Group | Group 1
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Eyebrow Position
Description: Position of eyebrow at the medial canthus relative to orbital rim
Time Frame: At time of evaluation
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1
Number analyzed (Participants) | 40
mm | -3.22 (1.91)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No